CLINICAL TRIAL: NCT05790850
Title: Pre-Habilitation with Mindfulness and Exercise for Patients Undergoing Radical Cystectomy (PRIMER Trial)
Acronym: PRIMER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: American Cancer Society, Inc. (Other); Integrated Translational Health Research Institute of Virginia (iTHRIV) (Unknown)
Responsible Party: Principal Investigator, Christine Ibilibor, MD, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR210502
Record Dates: First submitted 2023-03-16; First posted 2023-03-30 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer; Non-muscle-invasive Bladder Cancer; Muscle-Invasive Bladder Carcinoma
Keywords: Mindfulness; Meditation; Physical Exercise; Pre-habilitation
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Usual preoperative care prior to radical cystectomy
- Intervention (Experimental): Preoperative pre-habilitation
  Interventions: Behavioral: Pre-operative physical exercise; Behavioral: Pre-operative mindfulness meditation practice

INTERVENTIONS:
Behavioral: Pre-operative physical exercise — Virtual instructor-guided twice weekly cycling-based high-intensity aerobic exercise program for a total of 30 days. Participants will use a study provided recumbent exercise bike and wristband fitness tracker to exercise and log the number of days they exercise with an instructor and self-directed cycling.
  Arms: Intervention
Behavioral: Pre-operative mindfulness meditation practice — Daily self-directed mindfulness practice involving a guided imagery meditation for a total of 30 days. Participants will use a study provided guided-imagery meditation audio file loaded to a study provided wristband fitness tracker. Participants will log the number of days they listen to the audio file or participate in self-directed solitary psychological support.
  Arms: Intervention

SUMMARY:
The PRIMER (Pre-Habilitation With Mindfulness and Exercise for Patients Undergoing Radical Cystectomy) trial is a pilot designed to estimate the feasibility of integrating a home-based pre-operative exercise and mindfulness program (pre-habilitation program) for patients scheduled to undergo radical cystectomy for bladder cancer in an attempt to improve both physical and psychological conditioning pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged ≥18 years of age
* Good surgical candidate determined by treating surgeon
* Histologically documented muscle invasive urothelial carcinoma of the bladder, high-risk non-muscle invasive bladder cancer, non-muscle invasive bladder cancer refractory to BCG, cisplatin ineligible muscle invasive bladder cancer receiving upfront cystectomy, urothelial carcinoma of the bladder with variant histology
* Adequate Organ Function per protocol definition
* ECOG performance status ≤2
* Received medical clearance to complete cardiopulmonary exercise testing
* Willing to use the personal or study provided devices for monitoring and performing the exercise routines.
* Fluent in English or Spanish for the EORTC QLQ questionnaire
* No known contraindications to high intensity exercise

Exclusion Criteria:

* Contraindications to participating in aerobic exercise
* Currently participating in an aerobic exercise program
* New onset chest pain nor dyspnea with exertion
* Histologically documented micropapillary or sarcomatoid bladder cancer
* Distant metastatic carcinoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patient-reported days devoted to solitary psychological support | 30 days
  Patient-reported days devoted to self-directed solitary psychological support related to cancer treatment during a 30 day period pre-operatively in the pre-habilitation program group
Number of patient-reported days devoted to exercise | 30 days
  Patient-reported minutes per day devoted to high-intensity exercise during a 30 day period pre-operatively in the pre-habilitation program group

SECONDARY OUTCOMES:
Post-operative complication rate | 30 days post-operatively
  Percentage of patients with a Clavien Grade 3 or higher complications at 30-days post-operatively
Patient-reported health-related quality of life as assessed by the European Organization for Research and Treatment of Cancer (EORTC) questionnaire. | 4-8 weeks pre-operatively, 2 weeks pre-operatively, 30 days post-operatively
  The EORTC QLQ BLM 30 consists of 30 questions developed to assess the quality of life of cancer patients. It incorporates nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale. Several single-item symptom measures commonly reported by cancer patients (dyspnea, loss of appetite, insomnia, constipation and diarrhea) and perceived financial impact of the disease. The questionnaire was designed to be cancer-specific, multidimensional in structure, appropriate for self-administration, and applicable across a range of cultural settings. All of the scales and single-item measures range in score from 0 to 100. A higher score represents higher symptomatology in each respective domain.
Peak oxygen uptake as measured on cardiopulmonary exercise testing (CPET) | 4-8 weeks pre-operatively, 2 weeks pre-operatively, 30 days post-operatively
  Maximal oxygen uptake will be measured using a cycle ergometer-based cardiopulmonary exercise testing (CPET).
Dispositional mindfulness as assessed by the Mindfulness Awareness Attention Scale (MAAS) | 4-8 weeks pre-operatively, 2 weeks pre-operatively, 30 days post-operatively
  The Mindfulness Awareness Attention Scale (MAAS) is a 15-item scale designed to assess a core characteristic of mindfulness, namely, a receptive state of mind in which attention, informed by a sensitive awareness of what is occurring in the present, simply observes what is taking place. Total scores range from 0 to 6; higher scores indicate higher dispositional mindfulness.
Perceived stress as assessed by the Perceived Stress Scale 10 (PSS 10) | 4-8 weeks pre-operatively, 2 weeks pre-operatively, 30 days post-operatively
  the Perceived Stress Scale 10 (PSS 10) is a 10-item survey that captures the respondent's stress level in the past month and uses a Likert scale to assess different domains of stress. Individual scores on the PSS 10 can range from 0 to 40 with higher scores indicating higher perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Summary of trial outcome data through publication or grant reporting requirements.